CLINICAL TRIAL: NCT03352167
Title: Antibiotic Resistance in Danish Emergency Departments. Prevalence, Risk Factors and Definition of Risk Groups.
Brief Title: Antibiotic Resistance in Danish EDs.
Acronym: AB-RED
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Christian Backer Mogensen, ass. professor, University of Southern Denmark
Other Study IDs: SHS-ED-11-2017
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Antibiotic Resistance, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Biospecimen Retention: Samples With DNA — swabs from nose, throat and rectum for analysis of bacterial DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- ED Hjoerring
- ED Aalborg
- ED Aarhus
- ED Herning
- ED Aabenraa
- ED Odense
- ED Slagelse
- ED Koege

SUMMARY:
The spread of multiresistant bacteria is an increasing problem which will mean increased costs, morbidity and mortality in the coming years. Emergency departments (ED) play a key role in the early identification and management of patients who are carriers of multiresistant bacteria, but today there is very limited knowledge about both prevalence in the EDs and risk factors for the carrier status of methicillin resistant Staphylococcus aureus (MRSA), extended spectrum beta lactam producing enterobacteria (ESBL), vancomycin resistant enterococci (VRE), carbapenem resistant enterobacteria (CPE) and toxin-producing Clostridium difficile (CD). This knowledge is necessary to prioritize and target the preventive response to the spread of multiresistant bacteria.

The aim of this project is to provide a comprehensive overview of prevalence and risk factors for carrier status at a national level, and to develop screening tools for early identification of MRSA, ESBL, VRE, CPE and CD carriers among patients admitted to Danish emergency departments.

For hospitalized patients in 8 emergency departments in 4 Danish regions, a total of 10,600 patients are asked for possible risk factors for resistant bacterial carrier status, and are swabbed in the throat, nose and rectum openings and examined for MRSA, VRE, CPE, ESBL and CD with the same analytical method of 4 clinical microbiological departments.

The results are analyzed so that the prevalence of resistant bacteria can be described at the hospital level, regional level and national level. Risk factors are analyzed for applicability for carrier identification, and based on this, screening models for the identification of carriers are developed.

The vision for the project is that, based on the collected data, a comprehensive picture of the extent of the problem in Denmark can be drawn up and new screening tools for early identification of carriers can be developed so that the intra-hospital spread of resistant bacteria can be met through early intervention with infectious hygiene measures.

The project has been granted a grant of DKK 3,000,000 from the Ministry of Health and the Elderly on December 7, 2016 and DKK 554,871 from the Region of Southern Denmark on 28 August 2017.

ELIGIBILITY:
* Must be over 18 years
* Must be admitted to one of the emergency departments selected for the project for more than 4 hours.
* Must be mentally competent
* To consent to participate

Exclusion Criteria:

* admitted more than 16 hours before inclusion
* no operation in rectum less than 2 weeks before the admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients more than 18 years of age admitted for any reason to one of the participating Emergency Departments
Sampling Method: Non-Probability Sample
Enrollment: 5117 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Bacterial Antibiotic Resistance | baseline observation only

CONTACTS AND LOCATIONS:
Locations (8):
- Denmark (8):
  - Hospital of Southern Jutland, Aabenraa
  - Aalborg University Hospital, Aalborg
  - Aarhus Univerisity Hospital, Aarhus
  - Herning Hospital, Herning
  - Hjørring Hospital, Hjørring
  - Køge University Hospital, Køge
  - Odense University Hospital, Odense
  - Slagelse Hospital, Slagelse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skjot-Arkil H, Mogensen CB, Lassen AT, Johansen IS, Chen M, Petersen P, Andersen KV, Ellermann-Eriksen S, Moller JM, Ludwig M, Fuglsang-Damgaard D, Nielsen FE, Petersen DB, Jensen US, Rosenvinge FS. Carrier prevalence and risk factors for colonisation of multiresistant bacteria in Danish emergency departments: a cross-sectional survey. BMJ Open. 2019 Jun 27;9(6):e029000. doi: 10.1136/bmjopen-2019-029000. PMID 31253624
- [Derived] Mogensen CB, Skjot-Arkil H, Lassen AT, Johansen IS, Chen M, Petersen P, Andersen KV, Ellermann-Eriksen S, Moller JM, Ludwig M, Fuglsang-Damgaard D, Nielsen F, Petersen DB, Jensen US, Rosenvinge FS. Cross sectional study of multiresistant bacteria in Danish emergency departments: prevalence, patterns and risk factors for colonization (AB-RED project). BMC Emerg Med. 2018 Aug 20;18(1):25. doi: 10.1186/s12873-018-0178-1. PMID 30126361